CLINICAL TRIAL: NCT02380521
Title: Effect of Exenatide Once Weekly on Cardiovascular Risk Markers in Patients With Type-2 Diabetes
Brief Title: Exenatide Once Weekly, Cardiovascular Risk and Type-2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Palermo (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Principal Investigator, Manfredi Rizzo, Associate Professor, University of Palermo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ESR-14-10139
Record Dates: First submitted 2015-02-15; First posted 2015-03-05 (Estimated); Last update posted 2016-11-08 (Estimated); Status verified 2016-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Exenatide once weekly; T2DM; IMT; Atherogenic lipoproteins
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Exenatide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 60 patients with T2DM (Experimental): These patients will be treated with exenatide once weekly for a period of 8 months
  Interventions: Drug: Exenatide once weekly (BYDUREON™)

INTERVENTIONS:
Drug: Exenatide once weekly (BYDUREON™) — Exenatide is considered investigational medicinal product (IMP) and will be prescribed to enrolled patients in accordance with local requirements.
  Exenatide will be available at a fixed dose of 2 mg and supplied as a kit. Exenatide should be injected subcutaneously (SC) in the thigh, upper arm (deltoid region) or abdomen. The injection site does not have to be consistent throughout the study. Injection can be done at any time of the day irrespective of meals. It is recommended that the time of injection is consistent throughout the study. Subjects will be instructed to perform an air shot before the first injection.
  Subjects will follow a fixed dose of 2 mg
  Other Names: BYDUREON™

SUMMARY:
The glucagon-like peptide 1 (GLP-1) agonist exenatide represents an effective therapy in patients with type 2 diabetes mellitus (T2DM), which also seems to have some important non-glycemic effects. Yet, these non-glycemic effects are still largely unknown.

The effect of exenatide once weekly was investigated in controlled, blinded and open-label clinical studies in subjects with T2DM who were controlled on diet and exercise alone or in combination with oral antidiabetic agents, but also in multi-dose controlled studies and such studies resulted in significant reductions in glycemic parameters (mean glycated hemoglobin (HbA1c), fasting serum/plasma glucose as well as postprandial plasma glucose levels), but also in body weight, over 24 to 30 weeks. Meaningful reductions were observed as early as week 4 of treatment, and maintained through 6 years of treatment.

The study investigating cardiovascular effects of exenatide once weekly is currently undergoing. The results available are not numerous (such as DURATION-2, DURATION-3, DURATION-4 studies) and cannot lead to definitive conclusions.

In this study the investigators will evaluate the effect of exenatide once-weekly on multiple cardiovascular risk markers. These markers are related to subclinical atherosclerosis, endothelial dysfunction, oxidative stress and atherogenic lipoproteins.

The investigators will perform an open label, single-arm, prospective, intervention study using exenatide once weekly for a period of 8 months on 60 patients with T2DM.

DETAILED DESCRIPTION:
The research hypothesis is to assess whether exenatide once weekly can reduce subclinical atherosclerosis (as measured by carotid-intima media thickness [cIMT]) in patients with T2DM.

The primary objective is to assess whether exenatide once weekly can reduce subclinical atherosclerosis (as measured by cIMT) in patients with T2DM.

Primary endpoint: Reduction in cIMT. The secondary objective is to assess whether exenatide once weekly can reduce atherogenic lipoproteins, oxidative stress and endothelial dysfunction in patients with T2DM.

Secondary endpoint: Reduction in atherogenic lipoproteins, oxidative stress and improvement of endothelial dysfunction.

The purpose of the present 8 months study is to elucidate largely unknown non-glycemic effects of exenatide as add-on to metformin, including effects on cIMT, oxidative stress parameters and atherogenic lipoproteins, in addition to its benefit on glycemic control, weight loss and other efficacy parameters, as well as the safety profile of exenatide.

The data for clinical and biochemical analyses, including collection of efficacy variables, ECG, pulse and physical examination, will be collected at baseline and after 8 months of therapy (at 6 months of the treatment, only the routine laboratory analyses, including HbA1c, will be performed).

Clinical diagnostic tools will include the measurement of:

1. cIMT, that will be assessed by B-mode real-time ultrasound using a single sonographer (Medison SonoAce Pico, with a probe of 7.5-10.0 MHz) in a standardized manner with fixed angles of insonation;
2. Endothelial dysfunction, that will be assessed by flow mediated dilation of brachial artery.

Biochemical analyses will include the analysis of:

1. Routine testing: blood testing, liver and kidney profile, plasma lipids, glucose metabolism parameters;
2. Oxidative stress parameters (plasma glutathione, serum lipid hydroperoxides, reactive oxygen species);
3. Atherogenic lipoproteins, e.g. the analysis of 11 distinct lipoproteins including very-low-density lipoprotein (VLDL), 3 intermediate density lipoprotein (IDL) subclasses and 7 low density lipoprotein (LDL) subclasses.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of informed consent prior to any study specific procedures;
2. Men and women with T2DM aged >18 years;
3. BMI >25 kg/m2;
4. HbA1c 7.5-8.5 %;
5. Receiving metformin therapy (doses ranging from 1500 to 3000 mg daily) for at least 8 weeks.

Exclusion Criteria:

1. Pregnancy or willingness to become pregnant;
2. Moderate and severe liver dysfunction;
3. Moderate and severe renal failure;
4. Previous major cardiovascular event;
5. Severe infections at the discretion of the investigator (such as human immunodeficiency virus [HIV], hepatitis B virus [HBV] and hepatitis C virus [HCV]);
6. Any malignancy;
7. Plasma triglycerides >400 mg/dL, plasma LDL-cholesterol > 250 mg/dL.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2016-07 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Subclinical atherosclerosis (as measured by cIMT) in patients with T2DM treated with exenatide once weekly | Change from baseline to 8 months of the treatment
  Reduction in cIMT after 8 months of the treatment

SECONDARY OUTCOMES:
Atherogenic lipoproteins (as measured by the analysis of 11 distinct lipoprotein subclasses using the Lipoprint system®) in patients with T2DM treated with exenatide once weekly | Change from baseline to 8 months of the treatment
  Reduction in atherogenic lipoproteins including small dense LDL particles after 8 months of the treatment
Oxidative stress (as measured by markers of oxidative stress) in patients with T2DM treated with exenatide once weekly | Change from baseline to 8 months of the treatment
  Reduction in oxidative stress after 8 months of the treatment
Endothelial dysfunction (as measured by flow mediated dilation of brachial artery) in patients with T2DM treated with exenatide once weekly | Change from baseline to 8 months of the treatment
  Improvement of endothelial dysfunction as indicated by changes in flow mediated dilation of brachial artery after 8 months of the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Montalto, MD, Study Director — University of Palermo
Locations (1):
- University Hospital of Palermo, Palermo, Italy

REFERENCES:
- [Background] Drucker DJ, Buse JB, Taylor K, Kendall DM, Trautmann M, Zhuang D, Porter L; DURATION-1 Study Group. Exenatide once weekly versus twice daily for the treatment of type 2 diabetes: a randomised, open-label, non-inferiority study. Lancet. 2008 Oct 4;372(9645):1240-50. doi: 10.1016/S0140-6736(08)61206-4. Epub 2008 Sep 7. PMID 18782641
- [Background] Bergenstal RM, Wysham C, Macconell L, Malloy J, Walsh B, Yan P, Wilhelm K, Malone J, Porter LE; DURATION-2 Study Group. Efficacy and safety of exenatide once weekly versus sitagliptin or pioglitazone as an adjunct to metformin for treatment of type 2 diabetes (DURATION-2): a randomised trial. Lancet. 2010 Aug 7;376(9739):431-9. doi: 10.1016/S0140-6736(10)60590-9. Epub 2010 Jun 26. PMID 20580422
- [Background] Diamant M, Van Gaal L, Stranks S, Northrup J, Cao D, Taylor K, Trautmann M. Once weekly exenatide compared with insulin glargine titrated to target in patients with type 2 diabetes (DURATION-3): an open-label randomised trial. Lancet. 2010 Jun 26;375(9733):2234-43. doi: 10.1016/S0140-6736(10)60406-0. PMID 20609969
- [Background] Russell-Jones D, Cuddihy RM, Hanefeld M, Kumar A, Gonzalez JG, Chan M, Wolka AM, Boardman MK; DURATION-4 Study Group. Efficacy and safety of exenatide once weekly versus metformin, pioglitazone, and sitagliptin used as monotherapy in drug-naive patients with type 2 diabetes (DURATION-4): a 26-week double-blind study. Diabetes Care. 2012 Feb;35(2):252-8. doi: 10.2337/dc11-1107. Epub 2011 Dec 30. PMID 22210563
- [Background] Blevins T, Pullman J, Malloy J, Yan P, Taylor K, Schulteis C, Trautmann M, Porter L. DURATION-5: exenatide once weekly resulted in greater improvements in glycemic control compared with exenatide twice daily in patients with type 2 diabetes. J Clin Endocrinol Metab. 2011 May;96(5):1301-10. doi: 10.1210/jc.2010-2081. Epub 2011 Feb 9. PMID 21307137
- [Background] Buse JB, Nauck M, Forst T, Sheu WH, Shenouda SK, Heilmann CR, Hoogwerf BJ, Gao A, Boardman MK, Fineman M, Porter L, Schernthaner G. Exenatide once weekly versus liraglutide once daily in patients with type 2 diabetes (DURATION-6): a randomised, open-label study. Lancet. 2013 Jan 12;381(9861):117-24. doi: 10.1016/S0140-6736(12)61267-7. Epub 2012 Nov 7. PMID 23141817